CLINICAL TRIAL: NCT06037915
Title: Airway Interventions During Intravenous Anesthesia in Children Undergoing Direct Laryngoscopy for Surgical Procedures Using High Flow Nasal Versus Low Flow Oxygen. A Pilot Study.
Brief Title: Airway Interventions During Intravenous Anesthesia in Children Undergoing Direct Laryngoscopy for Surgical Procedures Using High Flow Nasal Versus Low Flow Oxygen. A Pilot Study.(Flowkid)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 003125
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Laryngoscopy; Child; Oxygen Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low flow oxygen (Active Comparator)
  Interventions: Device: low flow oxygen with nasopharyngeal tube
- high flow oxygen (Active Comparator)
  Interventions: Device: high flow oxygen with OptiflowTM Nasal High Flow

INTERVENTIONS:
Device: low flow oxygen with nasopharyngeal tube — low flow oxygen with nasopharyngeal tube
  Arms: low flow oxygen
Device: high flow oxygen with OptiflowTM Nasal High Flow — high flow oxygen with OptiflowTM Nasal High Flow
  Arms: high flow oxygen

SUMMARY:
The goal of this clinical trial is to evaluate possible differences in airway responses and interventions during intravenous anesthesia for direct laryngoscopy in children when comparing two oxygenation methods (conventional low flow oxygen supplementation via nasopharyngeal tube versus Nasal High Flow Therapy with the OptiflowTM system ).

DETAILED DESCRIPTION:
Surgical procedures during direct laryngoscopy is performed under general anesthesia with spontaneous or controlled ventilation. These therapeutic procedures, such as the supraglottoplasty, are a challenge for both the surgeon and the anesthesiologist. While the airway should be freely accessible for the surgeon, the main concern of the anesthesiologist is adequate sedation, preservation of the free airway and oxygenation. Prevention of under-or over-sedation, with careful titration of sedation according to patient needs and preservation of spontaneous ventilation are challenging, especially in children.Traditionally low flow oxygen supplementation via nasopharyngeal tube was used for oxygenation during the surgery. However, it is known that 'in adults', the reported safe apnea time can be extended by using high flow nasal oxygen and this method is therefore increasingly used for oxygenation. Previous studies have already reported that the application of high-flow 100 percent(%) oxygen in children allowed for an apnea time of more than 7 minutes without desaturation. Interestingly, time to desaturation was not lowered when low-flow 100% oxygen via nasal cannula was used, compared to high flow oxygen.

The OptiflowTM Nasal High Flow (NHF) Therapy system (Fisher and Paykel Healthcare - Auckland New Zealand) is a form of non-invasive respiratory therapy (Fig.1). This system can deliver high levels of oxygen (FiO2 21% up to 100%). The higher flow rates provide a reduction of dead space and a dynamic, positive airway pressure, both of which can increase alveolar ventilation. A critical distinctive element of NHF therapy is airway hydration, i.e., heated humidification. Heating and humidifying not only makes high gas flows tolerable for patients but also prevents desiccation of the airway epithelium and maintains and improves mucociliary clearance.The Fisher & Paykel Healthcare Optiflow Junior 2 Nasal Interface is a non-sealing nasal interface specifically designed for the flow requirements and anatomical features of neonates, infants and children on NHF therapy.

In this trial, minor participants scheduled for elective direct laryngoscopy with surgical intervention will be enrolled, provided that they comply with in-and exclusioncriteria and that an informed consent was given by the parent or legal guardian. All included children will be premedicated with midazolam 0.05 mg/kg. Standard monitoring including 3-lead electrocardiography, non-invasive blood pressure, peripheral pulse-oximetry, respiratory rate and rectal temperature will be continuously monitored and recorded. To evaluate the depth of sedation, the NeuroSENSE ® monitor will be installed previous to anesthesia induction. After induction of anesthesia a 24 Gauge intravenous catheter is placed in a peripheral vein. Baseline parameters of heart rate and blood pressure will be noted at this timepoint. Induction of anesthesia will be carried out with sevoflurane and a bolus of dexmedetomidine of 4mcg/kg will be administered. Maintenance of anesthesia will be accomplished with dexmedetomidine infused at 2mcg/kg/h and adjusted to clinical needs with top up rate dexmedetomedine of 0.5 mcg/kg/h. Remifentanil will be infused at 0.3 mcg/kg/min and adjusted to clinical needs to 0.5 mcg/kg/min.Guidance of the titration of dexmedetomidine/remifentanil according to clinical signs, is standard of care. Before start of surgery, on visualizing the vocal cords, one spray of 10% Lidocaïne is delivered to anesthetize the vocal cords. The included participants will be randomized into two groups: low flow oxygen vs high flow nasal therapy. The REDCap randomization module will be used to randomize patients. According to randomization, children will receive Optiflow nasal prongs or nasal pharyngeal tube for oxygen supplementation. Spontaneous ventilation will be maintained. In case of laryngospasm and desaturation, propofol will be used as rescue medication. After surgery all children will be monitored on intensive care or PACU (Post Anesthetic Care Unit) as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective direct laryngoscopy with surgical intervention
* written informed consent of the parents or legal guardian

Exclusion Criteria:

* refusal of informed consent
* known allergy for dexmedetomidine
* known allergy for remifentanil
* pulse oxygen saturation (SpO2) is lower than 85%, at induction of anesthesia

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
the incidence of airway interventions | during surgery
  defined as the need to interrupt the procedure in order to maintain adequate oxygenation with mask ventilation, introduction of a nasopharyngeal airway or intubation with endotracheal tube
incidence of desaturation | during surgery
  defined as pulse oxygen saturation(SpO2) lower than 90% for more than 30 seconds
incidence of bradycardia | during surgery
  defined as a change of 30 percent beyond the baseline of heart rate
incidence of tachycardia | during surgery
  defined as a change of 30 percent beyond the baseline of heart rate

SECONDARY OUTCOMES:
Comparison of the oropharyngeal mucosa before and after the procedure | before induction of anesthesia and at end of surgery
  1= good quality, humid mucosa; 2= acceptable quality; 3= dry mucosa)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Aerts, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No